CLINICAL TRIAL: NCT07303985
Title: The Effects of Remimazolam on Cerebral Blood Flow Following General Anesthesia Induction
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Jun Zhang (Other)
Responsible Party: Sponsor-Investigator, Jun Zhang, Professor, Fudan University
Organization: Fudan University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2510-Exp296
Record Dates: First submitted 2025-12-12; First posted 2025-12-26 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Cerebral Blood Flow
Keywords: Remimazolam; Propofol; Cerebral blood flow
MeSH Terms: interventions — remimazolam; Propofol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Propofol (Other): Propofol is used as the sedative agent during the anesthesia induction period.
  Interventions: Drug: Propofol (Group P)
- Remimazolam (Experimental): Remimazolam is used as the sedative agent during the anesthesia induction period.
  Interventions: Drug: Remimazolam

INTERVENTIONS:
Drug: Remimazolam — Remimazolam is used as the sedative agent during the anesthesia induction period (administer remimazolam as an intravenous bolus of 0.3 mg/kg for induction).
  Other Names: Experimental
  Arms: Remimazolam
Drug: Propofol (Group P) — Propofol is used as the sedative agent during the anesthesia induction period (administer propofol at 2 mg/kg for induction).
  Other Names: Comparator
  Arms: Propofol

SUMMARY:
This study will enroll 40 subjects aged 18 years or older scheduled for elective surgery under general anesthesia with endotracheal intubation. Basic medical history information will be collected. Subjects will be divided into two groups of 20 each: a remimazolam group and a propofol group. The study period will span from one day before surgery to one day after surgery. The study will assess middle cerebral artery cerebral blood flow following general anesthesia induction and postoperative anesthesia recovery.

DETAILED DESCRIPTION:
A significant reduction in cerebral blood flow (CBF) frequently occurs following general anesthesia induction. This decrease in CBF can lead to a reduction in the delivery of oxygen and glucose to brain tissue. If the magnitude or duration of this reduction exceeds the compensatory capacity of cerebral autoregulation, it can result in an imbalance between cerebral oxygen supply and demand, thereby increasing the risk of cerebral ischemia and neurological injury. Patients who are elderly, have hypertension, a history of cerebrovascular disease (e.g., stroke, intracranial arterial stenosis), or pre-existing brain injury are at higher risk for pronounced CBF reduction after induction, making them more susceptible to postoperative cognitive dysfunction, exacerbation of existing deficits, or new ischemic events. This underscores the urgent need to identify effective and safe therapeutic strategies to mitigate this risk.

Remimazolam is a novel benzodiazepine agent, structurally derived from midazolam with the introduction of a metabolically labile methyl propionate side chain. It similarly acts on the GABAA receptor, promoting chloride ion influx and inhibiting neuronal electrical activity. Administered intravenously for sedation and hypnosis, it is characterized by rapid onset, short duration of action, rapid recovery, minimal accumulation, and metabolism independent of hepatic or renal pathways. Previous studies indicate that benzodiazepines generally lack significant cardiovascular depressant effects and are associated with a lower incidence of hemodynamic instability during anesthesia induction. However, the specific impact of remimazolam on CBF following general anesthesia induction remains unclear.

Therefore, to further elucidate the effects of this novel benzodiazepine, remimazolam-which reportedly lacks significant cardiovascular depression-on CBF post-induction, we propose the following strategies for our clinical study: (1) compare remimazolam with the commonly used agent propofol for anesthesia induction; (2) administer remimazolam as an intravenous bolus of 0.3 mg/kg and propofol at 2 mg/kg for induction; (3) implement goal-directed fluid management during the peri-induction period; (4) utilize ultrasound to monitor blood flow in the middle cerebral artery; and (5) assess postoperative recovery parameters. Through this comprehensive approach, we aim to determine whether remimazolam offers a protective or optimizing effect on CBF during general anesthesia induction, thereby providing an empirical foundation for its routine clinical use in this context.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have signed the informed consent form and are willing to comply with the study protoco
* Age greater than 18 years
* ASA physical status classification I to II
* Scheduled for elective surgery
* Undergoing general anesthesia with endotracheal intubation
* No history of cerebrovascular disease, carotid artery stenosis, or traumatic brain injury.

Exclusion Criteria:

* History of intracranial lesions, carotid artery stenosis, or traumatic brain injury
* Allergy or contraindications to remimazolam or propofol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Peak systolic blood flow velocity (PS) | 1, 3, 5, and 10 minutes after endotracheal intubation.
  Peak systolic blood flow velocity (PS) in the middle cerebral artery following general anesthesia induction (at 1, 3, 5, and 10 minutes after endotracheal intubation). Peak systolic blood flow velocity (PS) is the maximum speed of blood flow recorded during the systolic phase of the cardiac cycle, typically measured in centimeters per second (cm/s). Peak systolic blood flow velocity (PS) normal values are vessel-specific and age-dependent. In healthy adults, the commonly cited reference range for the middle cerebral artery (MCA) is approximately 80-120 cm/s. This value decreases with age. For other intracranial arteries, PS is generally lower (e.g., 40-80 cm/s for vertebrobasilar arteries). Physiological factors like hematocrit and gender also cause minor variations. Clinically, PS values above 140-200 cm/s in the MCA often indicate significant pathology such as vasospasm or stenosis.

SECONDARY OUTCOMES:
The resistance index (RI) of the middle cerebral artery | 1, 3, 5, and 10 minutes after endotracheal intubation
  The resistance index (RI) of the middle cerebral artery (MCA) is a hemodynamic parameter. It reflects downstream cerebrovascular resistance and is defined by the formula: RI = (Peak Systolic Velocity - End-Diastolic Velocity) / Peak Systolic Velocity.
  A normal RI in the MCA for healthy adults typically ranges from 0.50 to 0.70 (or 50-70%). Values are influenced by age, with neonates and infants having higher normal values (often up to 0.80-0.85) which decrease toward adult levels with maturation. In elderly individuals, a slight increase may be observed due to reduced vascular compliance.
  An elevated RI (>0.80) generally indicates increased distal vascular resistance, which can be caused by intracranial hypertension, severe microangiopathy, or brain death. A very low RI (<0.50) may suggest a hyperemic state or proximal stenosis.
Mean blood flow velocity (MV) | 1, 3, 5, and 10 minutes after endotracheal intubation
  Mean blood flow velocity (MV), often referred to as Time-Averaged Maximum Velocity (TAMV), is a key hemodynamic parameter measured by Doppler ultrasound. It represents the average speed of the fastest-moving blood cells within a vessel over one complete cardiac cycle.
  For the middle cerebral artery (MCA) in healthy adults, the normal MV typically ranges from 40 to 65 cm/s. This value is age-dependent, being higher in children and gradually decreasing with advancing age. A sustained MV outside this range, particularly when asymmetric compared to the contralateral side, can indicate pathological conditions such as stenosis, hyperemia, or impaired autoregulation. Its calculation integrates both systolic and diastolic flow, making it a stable indicator of overall cerebral perfusion.
Pulsatility index (PI) | 1, 3, 5, and 10 minutes after endotracheal intubation
  The Pulsatility Index (PI) is a dimensionless hemodynamic parameter derived from Transcranial Doppler (TCD) ultrasound. It quantifies the pulsatility of the blood flow waveform, reflecting downstream cerebrovascular resistance. It is calculated using the formula: PI = (Peak Systolic Velocity - End-Diastolic Velocity) / Mean Velocity.
  For the middle cerebral artery (MCA) in healthy adults, the normal PI typically ranges from 0.70 to 1.10. Age significantly influences this value; neonates have a much higher normal PI (often >1.50), which decreases to adult levels during childhood. An elevated PI (>1.20) generally indicates increased distal resistance, which can be caused by intracranial hypertension or small vessel disease. Conversely, a very low PI (<0.60) may suggest a hyperdynamic state or proximal stenosis.
Postoperative recovery time | During the post-anesthesia care unit (PACU)
  post-anesthesia care unit (PACU) length of stay. There is no single universal "normal value" for Post-Anesthesia Care Unit (PACU) length of stay, as it is highly dependent on the type of surgery, anesthesia technique, institutional protocols, and patient-specific factors. For straightforward, outpatient, or minor inpatient surgeries, a typical stay often ranges from 30 minutes to 2 hours. The primary discharge criteria are based on standardized scoring systems, most commonly the Aldrete score or its modifications. Patients must achieve a predetermined score (usually ≥9 out of 10) indicating stable vital signs, adequate oxygenation, intact consciousness, and controlled pain and nausea before discharge to a ward or home. Prolonged stays beyond expected benchmarks are used as a quality indicator to identify and address potential complications like postoperative nausea and vomiting, pain, or hemodynamic instability.
Postoperative cognitive score | On the first postoperative day.
  Postoperative cognitive score was assessed by the Mini-Mental State Examination, MMSE). MMSE is a standardized, 30-point questionnaire used to screen for cognitive impairment. It assesses five key domains: orientation (to time and place), registration and recall of words, attention and calculation (e.g., serial sevens), language abilities (naming, repetition, comprehension, reading, writing), and visual construction (copying a pentagon).
  Administration involves a trained examiner asking the patient specific questions in a quiet setting, typically taking 5-10 minutes. One point is awarded for each correct task, with a maximum total score of 30.
  Results are interpreted based on the total score: 27-30 suggests normal cognition, 24-26 indicates mild cognitive impairment, 19-23 signifies moderate impairment, and a score ≤18 points to severe impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Zhang, Principal Investigator — Fudan University Shanghai Cancer Centre
Locations (1):
- Fudan University Shanghai Cancer Centre, Shanghai, China

IPD SHARING:
Plan to Share IPD: No
The data sets are available from the corresponding author on reasonable request